CLINICAL TRIAL: NCT03446092
Title: A Pilot Investigation of a Mindfulness Course for People With Incurable Cancer
Brief Title: Mindfulness for People With Incurable Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster University (Other)
Collaborators: University Hospitals of Morecambe Bay NHS Trust (Other); Rosemere Cancer Foundation, UK (Unknown)
Responsible Party: Principal Investigator, Fiona Eccles, Lecturer, Lancaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRASProject ID: 226702
Record Dates: First submitted 2018-02-13; First posted 2018-02-26 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Cancer
Keywords: Cancer; Mindfulness; Palliative care
MeSH Terms: conditions — Neoplasms | interventions — Mindfulness; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness group (Experimental): Group will receive mindfulness intervention
  Interventions: Behavioral: Mindfulness for health

INTERVENTIONS:
Behavioral: Mindfulness for health — A course of mindfulness using the mindfulness for health programme.

SUMMARY:
The study will investigate whether a mindfulness course can help people with incurable cancer who are seen by oncologists in a particular National Health Service Hospital Trust in the United Kingdom.

DETAILED DESCRIPTION:
It can be hard to come to terms with living with a life limiting condition such as incurable cancer and individuals are at risk of experiencing high levels of psychological distress, which can often be overlooked when the focus is on managing physical symptoms.

Mindfulness-based interventions have been shown to be helpful in reducing distress for people with cancer generally. This pilot study will use an established mindfulness programme called mindfulness for health with people with cancer which is incurable to see if this type of intervention is acceptable and useful for this group of people.

ELIGIBILITY:
Inclusion Criteria:

* Deemed by the oncologist to have incurable cancer
* Patient of the University Hospitals of Morecambe Bay NHS Foundation Trust
* Treated by an oncologist
* Believe they are able to commit to attending most of the mindfulness course sessions
* Oncologist assesses they are well enough to participate in the intervention

Exclusion Criteria:

* Having any other condition or difficulty which the medical team thinks would compromise their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Acceptability and usefulness of intervention for participants | Within 4 weeks of the end of the intervention
  This will be a qualitative outcome, collected via semi-structured interview

SECONDARY OUTCOMES:
Acceptability and usefulness of intervention for participants- 3 months | 3 months following completion of the intervention
  This will be a qualitative outcome, collected via semi-structured interview
Change in depression anxiety and stress | Collected before the intervention (up to 4 weeks before the intervention) and within 4 weeks of the end of the intervention
  Using the Depression, Anxiety and Stress (DASS21) scale we will measure the change post intervention score - pre intervention score. Each subscale (depression, anxiety and stress) ranges from 0-21, with higher scores indicating higher distress. A greater decrease in scores, would mean a greater improvement in symptoms.
Change in depression anxiety and stress-3 months | Collected before the intervention (up to 4 weeks before the intervention) and 3 months after the end of the intervention
  Using the Depression, Anxiety and Stress (DASS21) scale we will measure the change post intervention score - pre intervention score. Each subscale (depression, anxiety and stress) ranges from 0-21, with higher scores indicating higher distress. A greater decrease in scores, would mean a greater improvement in symptoms.
Change in mindfulness | Collected before the intervention (up to 4 weeks before the intervention) and within 4 weeks of the end of the intervention
  Using the Five Factor Mindfulness Questionnaire we will measure pre-post change scores.
Change in mindfulness- 3 months | Collected before the intervention (up to 4 weeks before the intervention) and 3 months following the intervention
  Using the Five Factor Mindfulness Questionnaire we will measure pre-post change scores
Change in quality of life | Collected before the intervention (up to 4 weeks before the intervention) and within 4 weeks of the end of the intervention
  Using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire we will measure pre-post change scores
Change in quality of life - 3 months | Collected before the intervention (up to 4 weeks before the intervention) and 3 months following the intervention
  Using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire we will measure pre-post change scores

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Lancaster Infirmary, Lancaster, United Kingdom

IPD SHARING:
Plan to Share IPD: No